CLINICAL TRIAL: NCT01370395
Title: Assessment of Biomarkers for Diagnosis in Geriatric Patients With the Symptom of Chest Pain in the Emergency Room
Brief Title: Assessment of Biomarkers for Diagnosis in Geriatric Patients
Acronym: BOSCH1
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: Klinikum Nürnberg (Other)
Responsible Party: Principal Investigator, Philipp Bahrmann, MD, University of Erlangen-Nürnberg Medical School
Other Study IDs: BOSCH1
Record Dates: First submitted 2011-06-08; First posted 2011-06-09 (Estimated); Last update posted 2012-10-01 (Estimated); Status verified 2012-09

CONDITIONS: Acute Coronary Syndrome
Keywords: geriatrics; troponin; electrocardiography; diagnosis; myocardial infarction
MeSH Terms: conditions — Acute Coronary Syndrome; Disease; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and plasma blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Left ventricular function: According to the result of the echocardiographic exam, the patients will be divided into subgroups with (LV-EF>=55%) and without preserved ejection fraction (LV-EF<55%).

SUMMARY:
Elderly patients are often admitted to hospital because of chest pain that is atypical for angina pectoris. In case of inconclusive electrocardiograms, determination of troponin is important for the diagnosis of an acute coronary syndrome. A highly sensitive assay for troponin T has recently been developed, permitting measurements of concentrations that are lower by a factor 10 than those measureable with conventional assays. In patients with stable coronary artery disease these concentrations were significantly associated with the incidence of cardiovascular death and heart failure but not with myocardial infarction. Copeptin, a novel biomarker of endogenous stress, may improve the diagnostic performance of troponin for an acute coronary syndrome in elderly patients. Other biomarkers such as MR-pro-adrenomedullin and endothelin-1 could improve both the diagnostic and prognostic assessment of the physician in these patients.

DETAILED DESCRIPTION:
All patients admitted to the clinic of acute geriatric medicine during the first 6 months will be enrolled in the study. Included patients will be prospectively studied for cardiovascular events for a period of 24 months.

At admission, patient history, physical examination, prior medications, vital signs including heart rate, blood pressure, body temperature, and all comorbidities will be recorded by a physician. Blood samples will be collected at the time of presentation. Determination of regular laboratory values together with very low circulating troponin T, copeptin, MR-pro-adrenomedullin, ANP and endothelin-1 levels will be measured. An electrocardiogram will be taken in all patients at admission. An echocardiography measuring the function of the heart valves, left ventricular diameters, ejection fraction (LV-EF), and diastolic function will be performed in all patients by a cardiologist in order to differentiate other mechanisms for the release of troponin. According to the result of the echocardiographic exam, the patients will be divided into subgroups with (LV-EF>=55%) and without preserved ejection fraction (LV-EF<55%).

Objectives:

1. To investigate the incidence of acute coronary syndromes in geriatric patients by measurement of very low circulating troponin T and copeptin levels.
2. To determine cardiovascular events, including cardiovascular death, fatal and nonfatal heart failure, and fatal and nonfatal acute myocardial infarction, of these patients during 24 months.
3. To analyze the relationship between very low circulating troponin T and cardiovascular events in these patients.
4. To analyze risk factors in geriatric patients with elevated troponin T for cardiovascular events.
5. To analyze whether the combined measurement of troponin T and copeptin or other markers improves the sensitivity for identification of acute coronary syndromes in geriatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 70 or older
* Signed informed consent

Exclusion Criteria:

* Hospitalization for unstable angina pectoris within the last 2 month
* ST-segment elevation myocardial infarction
* Heart valve defects with need for surgical intervention
* Coronary bypass surgery or percutaneous transluminal angioplasty within the last 3 months
* Planned elective coronary revascularization
* Serum creatinine> 2.0 mg / dl (177 µmol / liter)
* Serum potassium> 5.5 mmol / l
* Limited survival probability within the next 3 months

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Emergency department of the Klinikum Nürnberg (50,000 attendances per year; the department caters to an urban population of approximately 1 million).
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2011-01; Primary Completion 2013-07 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
cardiovascular death | 24 months

SECONDARY OUTCOMES:
fatal and nonfatal acute myocardial infarction | 24 months
fatal and nonfatal heart failure | 24 months
  hospitalization for fatal and nonfatal heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Bahrmann, MD, Principal Investigator — Department of Internal Medicine II-2, Chair of Internal Medicine V, Institute for Biomedicine of Ageing, Friedrich-Alexander-Universität Erlangen-Nürnberg
Locations (1):
- Klinikum, Nuremberg, Germany

REFERENCES:
- [Derived] Bahrmann P, Christ M, Bahrmann A, Rittger H, Heppner HJ, Achenbach S, Bertsch T, Sieber CC. A 3-hour diagnostic algorithm for non-ST-elevation myocardial infarction using high-sensitivity cardiac troponin T in unselected older patients presenting to the emergency department. J Am Med Dir Assoc. 2013 Jun;14(6):409-16. doi: 10.1016/j.jamda.2012.12.005. Epub 2013 Jan 30. PMID 23375478
- [Derived] Bahrmann P, Bahrmann A, Breithardt OA, Daniel WG, Christ M, Sieber CC, Bertsch T. Additional diagnostic and prognostic value of copeptin ultra-sensitive for diagnosis of non-ST-elevation myocardial infarction in older patients presenting to the emergency department. Clin Chem Lab Med. 2013 Jun;51(6):1307-19. doi: 10.1515/cclm-2012-0401. PMID 23314553